CLINICAL TRIAL: NCT00743418
Title: The Use of Advanced Tracking Technologies for the Analysis of Mobility in Alzheimer's Disease and Related Cognitive Disorders
Brief Title: Tracking Technologies for the Analysis of Mobility in Alzheimer's Disease
Acronym: SenTra
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr' Jeremia Heinik, Psychogeriatric clinic, Sourasky Medical Center, Tel-Aviv Israel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DIP-K.3.1.
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2008-08-28 (Estimated); Status verified 2008-08

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Radio Frequency Identification Device

ARMS (3):
- 1 (Other): Healthy controls Mini Mental State evaluation score >28/30
  Interventions: Device: GPS modem and RFID
- 2 (Other): Mild Cognitive Impairment: Mini Mental State Evaluation Score (MMSE)=26-28/30
  Interventions: Device: GPS modem and RFID
- 3 (Other): Mild Dementia: Mini Mental State Evaluation Score (MMSE)=21-25/30
  Interventions: Device: GPS modem and RFID

INTERVENTIONS:
Device: GPS modem and RFID — The participant will take the GPS kit with him/her everywhere during the whole day for a period of 4 weeks. The GPS tracking kit consists of a GPS receiver with a GSM modem, an RF transmitter contained in a wrist-watch and a monitoring unit located in the home that enables researchers to know whenever the tracked person leaves home. The waterproof RF transmitter will allow researchers to know whether or not research subjects leave home with the GPS device and if they are carrying the device or not at a given moment.

SUMMARY:
The research is aimed at exploring the application of novel tracking technique for the study of spatial activity among dementia patients and its implication on their families. The study sample will be composed of three groups of volunteers, each including100 participants aged over 60 years. The first group will include MCI (Mild Cognitive Impairment) patients. The second group will include patients that suffer from mild dementia. The third group will include age matched healthy participants. The tracking equipment will be a GPS apparatus of 450 gms that will be carried by the participants for 24 hours along 2-4 weeks. The GPS data will be transferred via the cellular network to operator center at the Hebrew university at Jerusalem, and will be documented in assigned data files. This monitoring procedure will be held every year and along a period of five years. The impact of the patient behavior on the care giver will be studied by means of five interviews along the tracking period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MCI, Alzheimer's disease, or mixed type dementia; OR
* Healthy control subjects who meet the following criteria:

  * Mini Mental State (MMSE) of at least 21
  * Age 60 years or older
  * Patients with history of stroke which is not followed by cognitive decline may be included
  * Fluent language skills

Exclusion Criteria:

* Other dementias (e.g. vascular, frontotemporal, metabolic etc);
* Other major psychiatric disorders (e.g. major depression, schizophrenia);
* Substance abuse;
* MMSE 20 or less;
* Severe motor disturbances;
* Sensory deficits potentially affecting mobility; OR
* Severe physical disorders (e.g. cancer, major operation)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-06; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation tools include: Geriatric Depression Scale, functional health questionnaire (SF-36), Emotional well-being questionnaire (Positive and Negative Affect Schedule; PANAS), single Life Satisfaction question and the Zarit Burden Interview | Before and after interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Psychogeriatric clinic, Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Shoval N, Auslander GK, Freytag T, Landau R, Oswald F, Seidl U, Wahl HW, Werner S, Heinik J. The use of advanced tracking technologies for the analysis of mobility in Alzheimer's disease and related cognitive diseases. BMC Geriatr. 2008 Mar 26;8:7. doi: 10.1186/1471-2318-8-7. PMID 18366748